CLINICAL TRIAL: NCT06996860
Title: Acute Effect of Fascial Treatments on Performance in Adolescent Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: FİLİZ EYÜBOĞLU (Other)
Responsible Party: Sponsor-Investigator, FİLİZ EYÜBOĞLU, Dr. lecturer, Uskudar University
Organization: Uskudar University (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: USKUKAR UNIVERSİTY
Record Dates: First submitted 2025-05-04; First posted 2025-05-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Sports Physical Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- massage gun (Experimental): massage gun
  Interventions: Device: theragun
- foam roller (Experimental): foam roller
  Interventions: Device: foam roller
- general warm up (Experimental): general warm up
  Interventions: Other: general warm up

INTERVENTIONS:
Device: foam roller — fascial therapy for performance effect
  Arms: foam roller
Device: theragun — fascial therapy for performance effect
  Arms: massage gun
Other: general warm up — fascial therapy for performance effect
  Arms: general warm up

SUMMARY:
Acute effect of fascial applications on performance and flexibility in adolescent volleyball athletes.

DETAILED DESCRIPTION:
60 adolescent athletes aged between 13-20 will be included in the study to be carried out at Galatasaray Taç Sports Facilities. Athletes will be divided into three groups by randomization: foam roller group, percussive therapy group and control group. For flexibility before fascial applications are applied to athletes; sit-and-reach test for agility performance; agility T test for jumping performance; CMJ (Counter movement jump) test will be performed. The sit-reach test will be repeated twice and the farthest point the athlete can reach will be recorded. In the CMJ test, the athlete will make 3 jumps with 30-second intervals and the highest value will be recorded. The t test will be repeated times and the best performance will be recorded. All athletes will have a general warm-up on a vertical bike (Monark Peak Bike, Sweden) with 74 watts (1.5 kg, 50 rpm) for five minutes. The foam roller group will start applying the foam roller one minute after the general warm-up is completed, and this application will be applied bilaterally for 30 seconds, from distal to proximal and from proximal to distal, for the gastrocnemius, quadriceps, hamstrings and gluteals muscles, respectively. For foam roller application, low density foam rollers will be used. After the application, the athletes will be subjected to CMJ, T agility and sit-reach tests, respectively. The percussive therapy group will be applied by the physiotherapist one minute after the general warm-up is completed, and this application will be applied bilaterally for 30 seconds, from distal to proximal and from proximal to distal, for the gastrocnemius, quadriceps, hamstrings and gluteals muscles, respectively. Percussive therapy will be applied using the Hypervolt device (Hyperice, California, USA) at a frequency of 40 Hz (2nd level), with an amplitude of 12 mm and a soft cap. After the application, the athletes will be subjected to CMJ, T agility and sit-reach tests, respectively. For the control group, CMJ, T agility and sit-reach tests will be performed again after the general warm-up.

Criteria for inclusion of athletes in the study; It was determined as having been exercising regularly for the last three months, exercising at least eight hours a week, and not having a lower extremity injury or surgical operation that would affect the test results. In addition, care was taken to ensure that they did not have any diabetes, epilepsy, neurological or neuromuscular health problems that would prevent them from participating in the test protocols explained in the details of the study. Athletes will be asked not to engage in strenuous physical activities and not to consume food, drinks or alcohol containing caffeine or similar stimulants for at least 24 hours before the test sessions.

ELIGIBILITY:
Inclusion Criteria:

* Having been playing volleyball for at least 2 years
* Having been training for at least the last month
* Training at least 8-10 hours a week
* No health problems that may prevent participation in the test protocol

Exclusion Criteria:

* Having had a previous injury in the lower extremity
* Having a condition that causes acute or chronic pain in the lower extremity
* Having had a surgical operation on the lower extremity

Ages: 13 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 68 (Actual)
Dates: Start 2024-03-27 (Actual); Primary Completion 2024-04-23 (Actual); Study Completion 2024-04-23 (Actual)

PRIMARY OUTCOMES:
counter movement jump testi | 10 minutes
  The CMJ test is a reliable test that measures the athlete's lower limb strength and jumping performance.
sit and reach flexibility test | 10 minutes
  Although the sit and reach test is considered a general flexibility performance measurement method, it specifically measures the flexibility of the lower extremity and hamstring muscle groups.
modified T test | 10 minutes
  The modified T test consists of 4 contact points formed in a T-shape in an area 5m long and 5m wide.

CONTACTS AND LOCATIONS:
Locations (1):
- Galatasaray Taç Sport Facilities, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Beardsley C, Skarabot J. Effects of self-myofascial release: A systematic review. J Bodyw Mov Ther. 2015 Oct;19(4):747-58. doi: 10.1016/j.jbmt.2015.08.007. Epub 2015 Aug 28. PMID 26592233
- [Background] Beckett JR, Schneiker KT, Wallman KE, Dawson BT, Guelfi KJ. Effects of static stretching on repeated sprint and change of direction performance. Med Sci Sports Exerc. 2009 Feb;41(2):444-50. doi: 10.1249/MSS.0b013e3181867b95. PMID 19127179